CLINICAL TRIAL: NCT03759119
Title: Use of a Tummy Time Intervention and Parent Education in Infants Born Preterm: a Randomized Control Trial
Brief Title: Use of a Tummy Time Intervention and Parent Education in Infants Born Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Kathryn Martin, Dawn Drumm, PT Physical Therapist, University of Indianapolis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-2239
Record Dates: First submitted 2018-11-20; First posted 2018-11-29 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial using a pretest /posttest control group design to allow for comparison between an intervention group that receives tummy time and parent education and a standard of care group that receives parent education only
Who Masked: Investigator
Masking Description: Outcome assessor investigator will be masked to all medical diagnoses of the infant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tummy Time and Parent Education (Experimental): This group will receive tummy time and parent education and be encouraged to perform tummy time on their own. They will utilize the PT Pal application to record their tummy time adherence. The primary investigator performs the intervention to the participants two times a day for 10 minutes for 4 weeks.
  Interventions: Behavioral: Tummy time and parent education; Behavioral: Parent education only
- Parent education (No Intervention): This group will receive parent education only and utilize the PT Pal application to record their adherence. The primary caregiver will be encouraged to perform the same dosage of tummy time (2x/day, 10 minutes each, 4 weeks) and record their adherence on the PT Pal application.

INTERVENTIONS:
Behavioral: Tummy time and parent education — Participants will receive tummy time positioning while awake for 10 minutes two times a day. Physiological monitoring will be maintained throughout the entire intervention and the intervention will be adjusted if needed to maintain stability. Participants will also receive parent education on tummy time prior to the tummy time intervention. The primary investigator will perform the tummy time intervention. Participants will be encouraged to continue performing tummy time on their own and record their adherence via the PT Pal application.
  Other Names: Group 1
  Arms: Tummy Time and Parent Education
Behavioral: Parent education only — Participants will receive the same tummy time education as those in the intervention group and will be asked to continue the intervention on their own and record their adherence via the PT Pal application.
  Steps of the intervention for group 2 (standard care).
  * Complete educational session with primary investigator.
  * Adherence during the four-week intervention period will be measured remotely through the PT Pal® application.
  Other Names: Group 2
  Arms: Tummy Time and Parent Education

SUMMARY:
The purpose of this research study is to see if tummy time and parent education helps motor development among infants born preterm. Participants will be recruited from Ann and Robert H. Lurie Children's Hospital of Chicago neonatal intensive care unit.

DETAILED DESCRIPTION:
The purpose of this randomized control trial will be to investigate the effects of a tummy time intervention, as compared to standard care, on motor outcomes among premature infants over a four-week period. Additionally, the study will measure tummy time adherence rates between groups post intervention for an additional four weeks.

To meet this purpose, the following objectives will be addressed:

1. To determine if there will be a difference in motor outcome scores on the Test of Infant Motor Performance (TIMP) among infants born preterm and utilizing a tummy time intervention and parent education compared to those in the standard care group receiving parent education only.
2. To determine if there will be a difference in adherence rates (average minutes/day) between groups among infants born preterm utilizing a tummy time intervention and parent education compared to those in the standard care group receiving parent education only.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, participants must meet the following inclusion criteria:

* born premature (< 37 weeks' gestation),
* require medical care within Lurie Children's NICU, be between 35 and 44 weeks postmenstrual age.
* Primary parent must have a working mobile device.
* Participants must be English or Spanish speaking as primary language.

Exclusion criteria:

* primary parent does not having a working mobile device and
* Speaking a language other than English or Spanish.
* Unable to be placed in the prone position,
* Physiologically unstable for handling
* Orally intubated or have a tracheostomy

Ages: 35 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Test of Infant Motor Performance (TIMP) for motor outcome | Change in motor outcome will be measured at initiation and at 8 weeks. Each participant will be enrolled in the study for 8 weeks. The study is expected to be completed within 6 months.
  The TIMP is a functional motor scale for newborns, including those born premature, up to infants four months corrected age, and was specifically designed for use in neonatal intensive care units (Rose & Westcott, 2005).

SECONDARY OUTCOMES:
PT Pal Application: Adherence | Change in adherence will be measured at initiation and at 8 weeks. Each participant will be enrolled in the study for 8 weeks. The study is expected to be completed within 6 months.
  The PT Pal application will be utilized to generate information back to the PI on adherence with tummy time outcomes of the prescription recommendations and thus serves as an adherence component for both the intervention and the standard care group.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Martin, DHSc, Study Chair — University of Indianapolis
Locations (1):
- Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Bentzley JP, Coker-Bolt P, Moreau NG, Hope K, Ramakrishnan V, Brown T, Mulvihill D, Jenkins D. Kinematic measurement of 12-week head control correlates with 12-month neurodevelopment in preterm infants. Early Hum Dev. 2015 Feb;91(2):159-64. doi: 10.1016/j.earlhumdev.2015.01.001. Epub 2015 Jan 23. PMID 25621433
- [Background] Campbell SK, Hedeker D. Validity of the Test of Infant Motor Performance for discriminating among infants with varying risk for poor motor outcome. J Pediatr. 2001 Oct;139(4):546-51. doi: 10.1067/mpd.2001.117581. PMID 11598602
- [Background] Lekskulchai R, Cole J. Effect of a developmental program on motor performance in infants born preterm. Aust J Physiother. 2001;47(3):169-76. doi: 10.1016/s0004-9514(14)60264-6. PMID 11552873
- [Background] Oberg GK, Campbell SK, Girolami GL, Ustad T, Jorgensen L, Kaaresen PI. Study protocol: an early intervention program to improve motor outcome in preterm infants: a randomized controlled trial and a qualitative study of physiotherapy performance and parental experiences. BMC Pediatr. 2012 Feb 15;12:15. doi: 10.1186/1471-2431-12-15. PMID 22336194